CLINICAL TRIAL: NCT07098741
Title: Comparative Analysis of Different Physiotherapy Interventions on Anterior Pelvic Tilt in Subjects With Non-Specific Low Back Pain: A Randomized Controlled Trial
Brief Title: Comparing Different Physiotherapy Interventions on APT in Non Specific Low Back Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Orthopedic and General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NOGH/MahtabAhmedPhD/0125/005
Record Dates: First submitted 2025-07-19; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Anterior Pelvic Tilt; Low Back Pain
Keywords: physiotherapy interventions; Non specific low back pain; anterior pelvic tilt; low back pain treatment
MeSH Terms: conditions — Low Back Pain | interventions — Electric Stimulation Therapy; Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: participants divided into four groups three interventional groups one control group
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A (Experimental): Core stability exercises with electrotherapy group.
  Interventions: Other: Core stability exercises with electrotherapy
- Group B (Experimental): Soft tissue release with manual therapy and stretching group.
  Interventions: Other: Soft tissue release with manual therapy and stretching
- Group C (Experimental): Postural correction exercises with contrast therapy group.
  Interventions: Other: Postural correction exercises with contrast therapy
- Group D (Experimental): (Control group) combination of electrotherapy with stretching and flexibility exercises group.
  Interventions: Other: combination of electrotherapy with stretching and flexibility exercises

INTERVENTIONS:
Other: Core stability exercises with electrotherapy — electrotherapy modalities for pain control will be used and exercises strengthening abdominal core muscles will be applied in two phases.
  Arms: Group A
Other: Soft tissue release with manual therapy and stretching — Manual soft tissue release will be performed and then stretching of back muscles and thigh muscles will be added to treatemnet.
  Arms: Group B
Other: Postural correction exercises with contrast therapy — Hot and cold packs will be used one after other for 10-15mins and specific exercises which are designed to improve posture will be taught and performed
  Arms: Group C
Other: combination of electrotherapy with stretching and flexibility exercises — some pain reducing electrotherapy modality like TENS will be used and general stretching and flexibility exercises will be performed
  Arms: Group D

SUMMARY:
Anterior pelvic tilt (APT) is a prevalent postural deviation characterized by excessive forward rotation of the pelvis, often resulting in increased lumbar lordosis. This condition is frequently associated with non-specific low back pain (NSLBP), which affects a significant portion of the global population and poses substantial challenges for individuals' well-being and healthcare systems worldwide. NSLBP is a multifactorial condition with various etiological factors, including poor posture, muscle imbalances, sedentary lifestyle, and biomechanical abnormalities such as APT. Understanding and effectively managing APT in the context of NSLBP is crucial for reducing pain, improving functional capacity, and enhancing quality of life for affected individuals .

Despite the prevalence and clinical significance of APT in NSLBP, there is a lack of comprehensive research comparing the effectiveness of different therapeutic interventions. Various approaches have been proposed, including core stability exercises, soft tissue release with manual therapy, stretching and flexibility exercises, and postural correction exercises . However, the relative efficacy of these interventions remains uncertain, hindering evidence-based decision-making in clinical practice.

A variety of therapeutic interventions have been proposed for managing APT and NSLBP, aiming to address underlying biomechanical imbalances, improve musculoskeletal function, and alleviate pain. Core stability exercises, focused on strengthening the deep stabilizing muscles of the spine and pelvis, have shown promise in improving postural alignment and reducing NSLBP symptoms. Soft tissue release techniques, such as manual therapy and myofascial release, target tight and restricted muscles associated with APT, promoting relaxation and improved range of motion. Stretching and flexibility exercises aim to elongate tight musculature, particularly in the hip flexors and lumbar extensors, thereby reducing excessive pelvic tilt and alleviating NSLBP. Additionally, postural correction exercises focus on retraining optimal alignment and body mechanics, promoting a more neutral pelvic position and reducing strain on the lumbar spine.

DETAILED DESCRIPTION:
Anterior pelvic tilt (APT) is a prevalent postural deviation characterized by excessive forward rotation of the pelvis, often resulting in increased lumbar lordosis. This condition is frequently associated with non-specific low back pain (NSLBP), which affects a significant portion of the global population and poses substantial challenges for individuals' well-being and healthcare systems worldwide. NSLBP is a multifactorial condition with various etiological factors, including poor posture, muscle imbalances, sedentary lifestyle, and biomechanical abnormalities such as APT. Understanding and effectively managing APT in the context of NSLBP is crucial for reducing pain, improving functional capacity, and enhancing quality of life for affected individuals.

Despite the prevalence and clinical significance of APT in NSLBP, there is a lack of comprehensive research comparing the effectiveness of different therapeutic interventions. Various approaches have been proposed, including core stability exercises, soft tissue release with manual therapy, stretching and flexibility exercises, and postural correction exercises. However, the relative efficacy of these interventions remains uncertain, hindering evidence-based decision-making in clinical practice.

Therefore, this study aims to address this gap in the literature by conducting a randomized controlled trial (RCT) to compare the effectiveness of core stability exercises, soft tissue release with manual therapy, stretching and flexibility exercises, and postural correction exercises in individuals with APT and NSLBP. By rigorously evaluating these interventions and their impact on APT, pain levels, functional capacity, and quality of life, this research seeks to provide valuable insights for clinicians and researchers, informing the selection and implementation of optimal treatment strategies for individuals with APT-related NSLBP.

Etiology and Biomechanics of Anterior Pelvic Tilt: The development of APT is multifactorial, involving a complex interplay of musculoskeletal factors, including muscle imbalances, joint stiffness, ligamentous laxity, and postural habits. Biomechanically, APT alters the alignment of the spine and pelvis, leading to increased stress on lumbar structures such as the intervertebral discs, facet joints, and surrounding musculature. This malalignment can contribute to aberrant movement patterns, decreased stability, and eventually, the onset of NSLBP.

Therapeutic Interventions for Anterior Pelvic Tilt and Non-Specific Low Back Pain: A variety of therapeutic interventions have been proposed for managing APT and NSLBP, aiming to address underlying biomechanical imbalances, improve musculoskeletal function, and alleviate pain. Core stability exercises, focused on strengthening the deep stabilizing muscles of the spine and pelvis, have shown promise in improving postural alignment and reducing NSLBP symptoms. Soft tissue release techniques, such as manual therapy and myofascial release, target tight and restricted muscles associated with APT, promoting relaxation and improved range of motion. Stretching and flexibility exercises aim to elongate tight musculature, particularly in the hip flexors and lumbar extensors, thereby reducing excessive pelvic tilt and alleviating NSLBP. Additionally, postural correction exercises focus on retraining optimal alignment and body mechanics, promoting a more neutral pelvic position and reducing strain on the lumbar spine.

Non-specific low back pain (NSLBP) is costly and widespread. Its lifetime prevalence is 80% and raises healthcare costs. High fear avoidance and Kinesio phobia are related with it, which causes long-term workplace illness. Stability (or 'core stability') exercises can reduce pain and impairment and be an effective treatment. Despite being the most prevalent physiotherapy treatment in the UK, there is no compelling evidence for it. This systematic review update examines stabilization exercises for NSLBP treatment and compares them to other exercises. Stabilization exercises outperformed other treatments for long-term pain and impairment in meta-analysis. Clinically negligible differences existed between groups. No statistical or clinically meaningful difference was seen between workout methods. The study found substantial evidence that stabilization exercises are not more helpful than other dynamic exercises over time. The low heterogeneity and large number of high-quality studies at long-term follow-up support our current findings, and subsequent research is unlikely to change this conclusion.

PROBLEM STATEMENT The high prevalence of anterior pelvic tilt (APT) among individuals with non-specific low back pain (NSLBP) represents a significant challenge in clinical management, as APT is linked to biomechanical imbalances and increased stress on lumbar structures. Despite its recognized role in contributing to NSLBP, there is a critical lack of comprehensive research evaluating the effectiveness of various therapeutic interventions designed to address APT. Current treatment approaches, including core stability exercises, manual therapy, stretching, and postural correction, remain inadequately supported by empirical evidence regarding their efficacy in reducing APT, alleviating pain, and enhancing functional capacity. This uncertainty not only complicates clinical decision-making but also limits the ability of healthcare professionals to implement evidence-based strategies. Therefore, this study seeks to investigate and compare the effectiveness of different interventions for managing APT in individuals with NSLBP, ultimately aiming to inform best practices and improve patient outcomes in this vulnerable population as it aims to determine the most effective intervention among these modalities for reducing anterior pelvic tilt and improving pain levels, functional capacity, and quality of life in this population.

OBJECTIVES OF THE STUDY 4.1 PRIMAERY OBJECTIVE: To assess and compare different physiotherapy interventions, including postural correction with contrast therapy, soft tissue release with manual therapy and stretching, core stability exercises with electrotherapy, and a combination of electrotherapy with stretching and flexibility exercises for treatment of Anterior Pelvic Tilt in Subjects with Non-Specific Low Back Pain.

4.2 SPECIFIC OBJECTIVES:

1. To compare the effectiveness of different interventions in reducing anterior pelvic tilt in subjects with non-specific low back pain.
2. To evaluate and compare the effects of these interventions on functional capacity (Range of Motion & Strength) in subjects with non-specific low back pain.
3. To assess and compare the effects of these interventions on pain levels in subjects with non-specific low back pain.
4. To assess and compare the effects of these interventions on quality of life in subjects with non-specific low back pain
5. To provide evidence-based recommendations for the selection and implementation of the most effective intervention for managing anterior pelvic tilt and non-specific low back pain based on the study outcomes.

SCOPE OF STUDY The scope of this study is designed to evaluate the effectiveness of various therapeutic interventions in managing Anterior Pelvic Tilt (APT) and associated Non-Specific Low Back Pain (NSLBP). This research aims to fill significant gaps in existing literature by providing a comprehensive analysis of how different treatments can alleviate pain, improve functional capacity, and correct postural deviations in affected individuals.

This study will primarily focus on four specific intervention modalities: postural correction with contrast therapy, soft tissue release with manual therapy and stretching, core stability exercises with electrotherapy, and a combination of electrotherapy with stretching and flexibility exercises. Each of these has been chosen based on their prevalence in current therapeutic practices and their potential impact on the biomechanical and muscular factors contributing to APT and NSLBP. The research will be conducted using a randomized controlled trial (RCT) design, the gold standard for clinical studies, to ensure the reliability of the results. Participants will be randomly assigned to one of the four intervention groups, with each group receiving a specific type of therapeutic intervention. The study will include both male and female adults aged 20-40 who have been clinically diagnosed with NSLBP associated with APT. Key outcome measures will include changes in pelvic tilt angle, pain intensity, quality of life and functional capacity. These outcomes will be assessed using reliable and validated tools such as digital photography with MicroDiCom software, Numeric Pain Rating Scale (NPRS) for pain, SF-36 questionnaire for quality of life and the lumbar range of motion and muscle strength for functional capacity. Assessments will be conducted at baseline, mid of interventions and immediately post-intervention to evaluate the effects of the applied interventions.

The geographical scope will include participants from multiple clinical settings across urban and suburban areas to enhance the diversity of the sample and increase the generalizability of the study findings by collaboration with multiple healthcare professionals to refer patients with NSLBP to participate in this study. By encompassing a broad demographic, the research aims to delineate more clearly the effectiveness of each intervention across diverse population subsets. Through rigorous evaluation and a well-defined scope, this study aspires to contribute significantly to the body of knowledge on managing APT and NSLBP, offering evidence-based recommendations that can be integrated into clinical practice for improved patient outcomes.

6.1 Conceptual Framework of Study: The purpose of the proposed research is to evaluate and compare the effects of different physiotherapy modalities on individuals who are suffering from non-specific low back pain and anterior pelvic tilt. The research will concentrate on the impact that these modalities have on pain levels, functional ability, craniovertebral angle, balance, and overall quality of life. There will be a total of one hundred volunteers in this experimental study, and they will be split into four unique groups: Group A will participate in exercises that focus on core stability and will also include electrotherapy; Group B will undergo soft tissue release in addition to manual therapy and stretching; Group C will engage in exercises that focus on postural correction and will also include contrast therapy; and Group D, which will serve as the control group, will take part in a combination of electrotherapy, stretching, and flexibility exercises. The purpose of this study is to determine which physiotherapy intervention is shown to be the most successful in improving functional outcomes and quality of life for patients who suffer from myofascial pain syndrome and radiculopathy. This will be accomplished by analyzing the outcomes across all of these groups. The findings will give useful insights into the optimization of treatment options for this patient population, which will ultimately lead to an improvement in therapeutic approaches in clinical practice.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Age: Participants must be between 20 and 40 years old.
2. Gender: Both genders, Male and Female have equal chance of selection as participant in the study.
3. Diagnosis: Participants must have a confirmed diagnosis of non-specific low back pain (NSLBP), altered lumbar posture, restricted range of motion of lumbar spine due to muscular spasm etc., altered anterior pelvic tilt angle by a qualified healthcare professional, based on standardized diagnostic criteria (e.g., clinical examination, imaging studies).
4. Confirmation of Anterior Pelvic Tilt (APT): Participants exhibiting APT confirmed through physical assessment by a trained examiner. This confirmation will involve the use of standardized measures such as digital inclinometers or goniometers.
5. Severity: Participants should have mild to moderate symptoms of non-specific low back pain (NSLBP) specially pain, as determined by the assessing healthcare provider.
6. Physical Capability: Participants who are physically capable of performing the prescribed exercises and interventions without significant limitations.
7. Consent: Participants who provide informed consent to participate in the study after receiving detailed information about the study objectives, procedures, potential risks, and benefits.
8. Compliance: Participants who are willing and able to comply with the study procedures, including attending scheduled sessions, adhering to the intervention protocols, and completing required assessments.
9. No Concurrent Treatment: Participants who have not undergone any concurrent treatments specifically targeting APT or low back pain during the study period to avoid confounding effects.

EXCLUSION CRITERIA:

1. Trauma or Fracture: Individuals with a history of trauma or fracture around the pelvic and lumbar region, as this may significantly affect the participant's ability to perform the prescribed exercises and interventions and confound study outcomes.
2. Orthopedic or Neurological Surgery: Participants with a history of orthopedic or neurological surgery related to the pelvic or lumbar region, as this may impact the participant's musculoskeletal function and response to the interventions.
3. Malignancy: Individuals with a diagnosis of malignancy, as this may introduce confounding variables and complicate the interpretation of study outcomes.
4. Autoimmune Disorders: Participants with autoimmune disorders affecting musculoskeletal function, as these conditions may influence the participant's response to interventions and introduce variability in study outcomes.
5. Referred or Radiating Visceral Pains: Individuals experiencing referred or radiating visceral pains, as these symptoms may indicate underlying pathologies requiring specific treatment and may confound the assessment of APT and NSLBP.
6. Gait Abnormalities and Neurological Disorders: Participants with gait abnormalities or neurological disorders affecting musculoskeletal function, as these conditions may influence the participant's ability to perform exercises and interventions and confound study outcomes.
7. Congenital and Developmental Disorders: Individuals with congenital or developmental disorders affecting musculoskeletal function, as these conditions may introduce variability in study outcomes and complicate the interpretation of results.
8. Pregnancy: Pregnant individuals will be excluded from the study due to the potential risks associated with certain physiotherapy modalities and the need for specialized considerations in this population.
9. Contraindications: Participants with contraindications to specific physiotherapy modalities included in the study protocol (e.g., contraindications to electrotherapy) will be excluded to ensure participant safety.
10. Inability to Attend Sessions: Participants who are unable to attend scheduled physiotherapy sessions due to logistical constraints (e.g., transportation issues, scheduling conflicts) will be excluded.
11. Cognitive Impairment: Participants with significant cognitive impairment or communication difficulties that may impede their ability to understand and follow study instructions will be excluded.
12. Participation in Other Research: Participants who are currently participating in other research studies involving treatment interventions for MPS and/or radiculopathy will be excluded to avoid potential confounding effects on outcomes and treatment adherence.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-03-20 (Actual); Primary Completion 2025-08-10 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
APT angle | 4 weeks
  Anterior pelvic tilt angle will be assessed before, at mid and at end of interventions
Pain | 4weeks
  Pain severity will be assessed using Numeric Pain Rating Scale NPRS. NPRS measures the pain severity quantitatively having zero "0" as no pain at one end and "10" as the worst ever pain at the other end. Higher the score on NPRS, more severe the pain and vice versa.

SECONDARY OUTCOMES:
Balance | 4 weeks
  Balance will be assessed using Y balnace test

CONTACTS AND LOCATIONS:
Overall Officials: Mazhar ALI, Phd, Study Chair — National orhtopedic and general hospital
Locations (1):
- National Orthopedic & General Hospital, Chak Four Hundred Fifty-four, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Due to ethical concerns

REFERENCES:
- [Background] Tan BT. A correlation study of the relationship between flat foot with anterior pelvic tilt and sacroiliac joints dysfunction among undergraduate students: UTAR; 2022.
- [Background] Kahere M, Hlongwa M, Ginindza TG. A Scoping Review on the Epidemiology of Chronic Low Back Pain among Adults in Sub-Saharan Africa. Int J Environ Res Public Health. 2022 Mar 3;19(5):2964. doi: 10.3390/ijerph19052964. PMID 35270657
- [Background] Algarni FS. Comparison of Abdominal and Hip Abductor Activation Between Chronic Low Back Pain and Asymptomatic Individuals During Walking. Masters Abstracts International; 2010.
- [Background] Mavajian M, Fakhari Z, Naghdi S, Bagheri H, Jalaie S. A pilot study on the short-term effects of myofascial release and core stability exercises on balance in chronic low back pain. Auditory and Vestibular Research. 2020.
- [Background] Shariat A, Anastasio AT, Soheili S, Rostad M. Home-based fundamental approach to alleviate low back pain using myofascial release, stretching, and spinal musculature strengthening during the COVID-19 pandemic. Work. 2020;67(1):11-19. doi: 10.3233/WOR-203248. PMID 32955470
- [Background] Kim B, Yim J. Core Stability and Hip Exercises Improve Physical Function and Activity in Patients with Non-Specific Low Back Pain: A Randomized Controlled Trial. Tohoku J Exp Med. 2020 Jul;251(3):193-206. doi: 10.1620/tjem.251.193. PMID 32669487
- [Background] Weng LM, Zheng YL, Peng MS, Chang TT, Wu B, Wang XQ. A Bibliometric Analysis of Nonspecific Low Back Pain Research. Pain Res Manag. 2020 Mar 9;2020:5396734. doi: 10.1155/2020/5396734. eCollection 2020. PMID 32215136
- [Background] Morris P, Ali K, Merritt M, Pelletier J, Macedo LG. A systematic review of the role of inflammatory biomarkers in acute, subacute and chronic non-specific low back pain. BMC Musculoskelet Disord. 2020 Mar 3;21(1):142. doi: 10.1186/s12891-020-3154-3. PMID 32126991
- [Background] Kahere M, Ginindza T. The burden of non-specific chronic low back pain among adults in KwaZulu-Natal, South Africa: a protocol for a mixed-methods study. BMJ Open. 2020 Sep 1;10(9):e039554. doi: 10.1136/bmjopen-2020-039554. PMID 32873683
- [Background] Bramah C, Mendiguchia J, Dos'Santos T, Morin JB. Exploring the Role of Sprint Biomechanics in Hamstring Strain Injuries: A Current Opinion on Existing Concepts and Evidence. Sports Med. 2024 Apr;54(4):783-793. doi: 10.1007/s40279-023-01925-x. Epub 2023 Sep 19. PMID 37725240
- [Background] Nagy P. The Biomechanical Demands of Ballet: Implications for Performance Profiling and Injury Aetiology: Edge Hill University; 2021
- [Background] Shojaei I, Salt EG, Bazrgari B. A prospective study of lumbo-pelvic coordination in patients with non-chronic low back pain. J Biomech. 2020 Mar 26;102:109306. doi: 10.1016/j.jbiomech.2019.07.050. Epub 2019 Aug 7. PMID 31427092
- [Background] Smith BE, Littlewood C, May S. An update of stabilisation exercises for low back pain: a systematic review with meta-analysis. BMC Musculoskelet Disord. 2014 Dec 9;15:416. doi: 10.1186/1471-2474-15-416. PMID 25488399

DOCUMENTS (3):
  • Study Protocol (2025-03-20): https://cdn.clinicaltrials.gov/large-docs/41/NCT07098741/Prot_000.pdf
  • Statistical Analysis Plan (2025-03-20): https://cdn.clinicaltrials.gov/large-docs/41/NCT07098741/SAP_001.pdf
  • Informed Consent Form (2025-03-20): https://cdn.clinicaltrials.gov/large-docs/41/NCT07098741/ICF_002.pdf